CLINICAL TRIAL: NCT04566770
Title: A Randomized, Double-blind, Placebo -Controlled Phase IIb Clinical Trial to Evaluate the Safety and Immunogenicity of Ad5-nCoV in Person 6 Years of Age and Older and Those Who Have Previously Been Vaccinated With Ad5-EBOV
Brief Title: A Clinical Trial of A COVID-19 Vaccine Named Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CanSino Biologics Inc. (Industry)
Collaborators: Beijing Institute of Biotechnology (Other); Jiangsu Province Centers for Disease Control and Prevention (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: JSVCT093
Record Dates: First submitted 2020-09-22; First posted 2020-09-28 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: COVID-19
Keywords: COVID-19; Vaccine; Ad5; Safety; Immunogencity; SARS-CoV-2; Adenovirus Vector
MeSH Terms: conditions — COVID-19; Alzheimer Disease 5

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- MID A (Experimental): 20 participants(18-49), Ad5-nCoV , two doses, Intramuscular administration
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector)
- MID B (Placebo Comparator): 10 participants(18-49), Ad5-nCoV-placebo , two doses, Intramuscular administration
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) -placebo
- MIN A (Experimental): 100 participants(6-17), Ad5-nCoV , two doses, Intramuscular administration
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector)
- MIN B (Placebo Comparator): 50 participants(6-17), Ad5-nCoV-placebo , two doses, Intramuscular administration
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) -placebo
- OLD A (Experimental): 100 participants(56 years of age and above), Ad5-nCoV , two doses(Low dose), Intramuscular administration
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector)
- OLD B (Experimental): 100 participants(56 years of age and above), Ad5-nCoV , two doses(Middle dose), Intramuscular administration
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector)
- OLD C (Placebo Comparator): 50 participants(56 years of age and above), Ad5-nCoV-placebo , two doses, Intramuscular administration
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) -placebo
- EBOV A (Experimental): 34 participants, Ad5-nCoV , two doses, Intramuscular administration
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector)
- EBOV B (Placebo Comparator): 17 participants, Ad5-nCoV , two doses, Intramuscular administration
  Interventions: Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) -placebo

INTERVENTIONS:
Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) — Intramuscular other name:Ad5-nCoV
  Arms: EBOV A; MID A; MIN A; OLD A; OLD B
Biological: Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) -placebo — Intramuscular other name:Ad5-nCoV
  Arms: EBOV B; MID B; MIN B; OLD C

SUMMARY:
This study is a randomized, double-blind, placebo -controlled IIb clinical trial, in order to evaluate the safety and immunogenicity of Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector) in people 6 years old and above and .

DETAILED DESCRIPTION:
This is a phase IIb clinical trial to evaluate safety and immuogenicity of Ad5-nCoV developed by Cansino and Beijing Institute of Biotechnology in health people aged 6 years old and above.

The study will be double-blind, placebo-controlled trial with participants randomly allocated 2:1 to placebo and experimental vaccine .

The immunization schedule is two doses intramuscular injections (deltoid).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 55 years old in MID group; aged 6-17 years old in MIN group; aged 56 years and above in OLD group; aged in EBO group is not limited.
* Able to understand the content of informed consent and willing to sign the informed consent
* Able and willing to complete all the secluded study process during the whole 6 months study follow-up period.
* Negative in HIV diagnostic test.
* Negative in serum antibodies (IgG and IgM) screening of COVID-19.
* Axillary temperature ≤37.0°C.
* General good health as established by medical history and physical examination.

Exclusion Criteria:

* Family history of seizure, epilepsy, brain or mental disease
* Subject allergic to any component of the investigational vaccine, or a more severe allergic reaction and history of allergies in the past.
* Woman who is pregnant, breast-feeding or positive in β-HCG (human chorionic gonadotropin) pregnancy test (urine) on day of enrollment, or become pregnant during the next 6 months
* Any acute fever disease or infections.
* History of SARS
* Major congenital defects or not well-controlled chronic illness, such as asthma, diabetes, or thyroid disease.
* Serious cardiovascular diseases, such as arrhythmia, conduction block, myocardial infarction, severe hypertension without controllable drugs, etc.
* Hereditary angioneurotic edema or acquired angioneurotic edema Urticaria in last one year
* No spleen or functional spleen.
* Platelet disorder or other bleeding disorder may cause injection contraindication
* Faint at the sight of needles.
* Prior administration of immunodepressant or corticosteroids, antianaphylaxis treatment, cytotoxic treatment in last 6 months.
* Prior administration of blood products in last 4 months
* Prior administration of other research medicines in last 1 month
* Prior administration of attenuated vaccine in last 1 month
* Prior administration of inactivated vaccine in last 14 days
* Current anti-tuberculosis prophylaxis or therapy
* According to the judgement of investigator,various medical, psychological, social or other conditions, those could affect the subjects to sign informed consent.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2022-01-19 (Actual)

PRIMARY OUTCOMES:
Safety indexes of adverse reactions | within 14 days post each vaccination
  Occurrence of adverse reactions post vaccination
Immunogencity indexes of GMT | Day 28 post the second vaccination
  Evaluate the Geometric mean titer (GMT) of IgG antibody
Immunogencity indexes of neutralizing antibody | Day 28 post the second vaccination
  Evaluate the Geometric mean titer (GMT) of neutralizing antibody

SECONDARY OUTCOMES:
Safety indexes of adverse events | Day 0-7,0-14,0-28 post each vaccination
  Occurrence of adverse reactions post-vaccination
Safety indexes of Hematological examination measures（Hemoglobin, WBC） | pre-vaccination, day 4 post each vaccination
  Occurrence of abnormal changes of Hematological examination indexes(only fit for MID and sentinel group)
Safety indexes of Blood routine measures(ALT, AST) | pre-vaccination, day 4 post each vaccination
  Occurrence of abnormal changes of lBlood routine indexes (only fit for MID and sentinel group)
Safety indexes of SAE | Within 6 months post the second vaccination
  Occurrence of serious adverse events post-vaccination
Immunogencity indexes of GMT | Day 28 post the first vaccination, pre the second vaccination ,Month 6 post the second vaccination
  Evaluate the Geometric mean titer of IgG antibody
Immunogencity indexes of neutralizing antibody | Day 28 post the first vaccination, pre the second vaccination ,Month 6 post the second vaccination
  Evaluate the Geometric mean titer (GMT) of neutralizing antibody
Immunogencity indexes of cellular immune | Day 28 post the first vaccination, pre and day 28 post the second vaccination
  Number of cell-mediated immune response against SARS-CoV-2（IL-2）

CONTACTS AND LOCATIONS:
Overall Officials: Fengcai Zhu, MSD, Principal Investigator — Jiangsu Provincal Center for Disease Control and Prevention
Locations (1):
- Taixing City center for Disease Control and Prevention, Taizhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feng JL, Wang WJ, Jin PF, Zheng H, Jin LR, Xia X, Zhang XY, Li ZP, Li JX, Zhu FC. Comparison of antibody persistency through one year between one-dose and two-dose regimens of Ad5-nCoV vaccine for COVID-19. Hum Vaccin Immunother. 2023 Aug 1;19(2):2230760. doi: 10.1080/21645515.2023.2230760. PMID 37428653
- [Derived] Zhu F, Jin P, Zhu T, Wang W, Ye H, Pan H, Hou L, Li J, Wang X, Wu S, Wang Y, Gou J, Huang H, Wu H, Wang X, Chen W. Safety and Immunogenicity of a Recombinant Adenovirus Type-5-Vectored Coronavirus Disease 2019 (COVID-19) Vaccine With a Homologous Prime-Boost Regimen in Healthy Participants Aged >/=6 Years: A Randomized, Double-Blind, Placebo-Controlled, Phase 2b Trial. Clin Infect Dis. 2022 Aug 24;75(1):e783-e791. doi: 10.1093/cid/ciab845. PMID 34551104